CLINICAL TRIAL: NCT05389722
Title: A Phase 1, Parallel-group, 3-part, 2-period, Fixed-sequence, Crossover, Open-label, Nonrandomized, Drug-drug Interaction Study to Assess the Pharmacokinetics of CC-92480 (BMS-986348) After Coadministration With Rifampin and Itraconazole, and Pharmacokinetics of Digoxin and Rosuvastatin After Coadministration With CC-92480 in Healthy Participants
Brief Title: A Study to Assess the Drug Levels of CC-92480 After Coadministration With Rifampin and Itraconazole, and the Drug Levels of Digoxin and Rosuvastatin After Coadministration With CC-92480 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA057-002
Record Dates: First submitted 2022-05-20; First posted 2022-05-25 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Healthy Volunteers
Keywords: CC-92480; Healthy Volunteer; Pharmacokinetic
MeSH Terms: interventions — Rifampin; Itraconazole; Digoxin; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1 (Experimental)
  Interventions: Drug: CC-92480; Drug: Rifampin
- Part 2 (Experimental)
  Interventions: Drug: CC-92480; Drug: Itraconazole
- Part 3 (Experimental)
  Interventions: Drug: CC-92480; Drug: Digoxin; Drug: Rosuvastatin

INTERVENTIONS:
Drug: CC-92480 — Specified dose on specified days
  Other Names: BMS-986348
Drug: Rifampin — Specified dose on specified days
  Arms: Part 1
Drug: Itraconazole — Specified dose on specified days
  Arms: Part 2
Drug: Digoxin — Specified dose on specified days
  Arms: Part 3
Drug: Rosuvastatin — Specified dose on specified days
  Arms: Part 3

SUMMARY:
The purpose of this study is to evaluate the drug levels of CC-92480 after coadministration with rifampin and itraconazole and the drug levels of digoxin and rosuvastatin after coadministration with CC-92480 in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Must have a body mass index between 18 and 33 kg/m2 (inclusive)
* Adult female of nonchildbearing potential or male, any race or ethnicity, and in good health as determined by the medical history, physical exam, vital signs, 12-lead electrocardiogram, and clinical laboratory assessments

Exclusion Criteria:

* Any surgical or medical condition possibly affecting drug absorption, distribution, metabolism, and excretion
* Any major surgery within 4 weeks of the first dose administration
* History of drug abuse within 2 years of the first dose administration

Other protocol-defined inclusion/exclusion criteria apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-06-09 (Actual); Primary Completion 2022-11-12 (Actual); Study Completion 2022-11-12 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Up to 2 months
Time of maximum observed plasma concentration (Tmax) | Up to 2 months
Area under the plasma concentration-time curve from time zero to the time of the last quantifiable concentration (AUC(0-T)) | Up to 2 months

SECONDARY OUTCOMES:
Number of participants with adverse events (AEs) | Up to 3 months
Number of participants with physical examination findings | Up to 3 months
Number of participants with vital sign abnormalities | Up to 3 months
Number of participants with 12-lead electrocardiogram (ECG) abnormalities | Up to 3 months
Number of participants with clinical laboratory abnormalities | Up to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Covance Clinical Research Unit - Dallas, Dallas, Texas, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm